CLINICAL TRIAL: NCT02228603
Title: How to Enhance Physical Activity After Cardiac Rehabilitation? A Randomised Controlled Study Comparing Two Follow-up Training Exercise Programs
Brief Title: Exercise as a Life-long Medicine in Patients With Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Helse Nord-Trøndelag HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014/92
Record Dates: First submitted 2014-08-27; First posted 2014-08-29 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Cardiovascular Diseases; Myocardial Infarction; Angina (Stable)
Keywords: exercise therapy; rehabilitation
MeSH Terms: conditions — Cardiovascular Diseases; Myocardial Infarction; Angina, Stable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- high-intensity exercise (Experimental): community-based group program: weekly supervised high-intensity exercise training during 8 weeks, followed by group counselling every third month for 12 months
  Interventions: Behavioral: high-intensity exercise training
- web-based follow-up (Active Comparator): web-based follow-up program: home-based group will be followed up by mail and telephone calls the first 8 weeks, then every third month for 12 months
  Interventions: Behavioral: web-based follow-up program
- control (Other): control group will receive usual care: information about recommended physical activity and healthy lifestyle
  Interventions: Behavioral: usual care

INTERVENTIONS:
Behavioral: high-intensity exercise training
  Arms: high-intensity exercise
Behavioral: web-based follow-up program
  Arms: web-based follow-up
Behavioral: usual care
  Arms: control

SUMMARY:
Exercise training is a core component in cardiac rehabilitation. Exercise adherence is, however, low after rehabilitation and the transition from supervised to unsupervised exercise is problematic for many patients with coronary artery disease. Therefore, it is important to provide extended services to improve exercise adherence and healthy lifestyle changes.

The aim of this study is to assess the effect of a time-limited intervention following out-patient cardiac rehabilitation on exercise adherence and cardiovascular risk reduction.

ELIGIBILITY:
Inclusion Criteria:

* myocardial infarction, stable angina, heart surgery
* finished phase 2 cardiac rehabilitation
* clinically stable
* able to communicate in Norwegian
* able to do a maximal treadmill test

Exclusion Criteria:

* unstable angina
* serious cardiac arrhythmia
* serious heart valve insufficiency
* heart failure
* any contraindication for high intensity exercise training
* participation in other exercise study
* pregnancy
* cognitive impairment
* drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
change in peak oxygen uptake | 2 years
  measured during exercise on treadmill (MetaMax Cortex/Innocor)

SECONDARY OUTCOMES:
physical activity | 2 years
  assessed by accelerometer SenseWear Armband Pro
quality of life | 2 years
  assessed by MacNew Health-related quality of life questionnaire
depression | 2 years
  assessed by Hospital anxiety and depression scale (HAD)

CONTACTS AND LOCATIONS:
Overall Officials: Asbjørn Støylen, prof, Principal Investigator — Norwegian University of Science and Technology
Locations (2):
- Norway (2):
  - Levanger Hospital, Levanger
  - St Olavs Hospital, Trondheim